CLINICAL TRIAL: NCT01750736
Title: The Use of a Home Exercise Program to Augment a Manual Therapy Intervention: a Randomized Controlled Trial
Brief Title: Manual Therapy and Augmented Exercise for Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Des Moines University (Other)
Collaborators: Walsh University (Other); Youngstown State University (Other)
Responsible Party: Principal Investigator, Shannon Petersen, Associate Professor, Des Moines University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DMUPT-001
Record Dates: First submitted 2012-12-11; First posted 2012-12-17 (Estimated); Last update posted 2015-02-12 (Estimated); Status verified 2015-02

CONDITIONS: Neck Pain
Keywords: Augmented Exercise; Cervicalgia; Manual Therapy; Manipulation; Quantitative Sensory
MeSH Terms: conditions — Neck Pain | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Augmented Exercise and Manual Therapy (Experimental): Subjects will receive manual therapy according to clinical guidelines followed by instruction in a specific exercise to augment the specific manual treatment provided.
  Interventions: Other: Augmented Exercise and Manual Therapy
- General Exercise and Manual Therapy (Active Comparator): Subjects will receive manual therapy according to clinical guidelines followed by instruction in a general neck range of motion exercise.
  Interventions: Other: General Exercise and Manual Therapy

INTERVENTIONS:
Other: Augmented Exercise and Manual Therapy — Session 1 will include the manual therapy intervention to cervical and or thoracic regions. Subjects will perform the augmented exercise at home and at each data collection session.
  Other Names: Manipulation; Mobilization; Self-Mobilization
  Arms: Augmented Exercise and Manual Therapy
Other: General Exercise and Manual Therapy — Session 1 will include the manual therapy intervention to cervical and or thoracic regions. Subjects will perform general range of motion exercises for the neck at home and at each data collection session.
  Other Names: Manipulation; Mobilization; Self-Mobilization
  Arms: General Exercise and Manual Therapy

SUMMARY:
Manual therapy and exercise have shown to be beneficial for people with neck pain, however it is not clear how outcomes following a general exercise program compare to specific exercises intended to augment a specific manual/hands-on intervention. This study will compare outcomes following manual therapy and a specific exercise program with manual therapy and a general exercise program.

DETAILED DESCRIPTION:
The purpose of this study is to determine if specific neck exercises intended to augment specific manual therapy treatments result in better outcomes than standard neck exercises in people with neck pain. Clinical tests and measurements as well as patient questionnaires will be completed and compared between groups.

A secondary purpose is to determine if self report of activity is correlated with functional improvements. We hypothesize that a specifically applied home exercise that augments the effects of the manual therapy intervention will lead to improvements in outcomes in patients with neck pain. We hypothesize that higher reports of self activity will be correlated with improvements in outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with complaint of neck pain, neck motion limitations, pain at end-range neck ROM, limited cervical/cervical and thoracic joint mobility, neck pain with manual segmental examination

Exclusion Criteria:

* The presence of any red flags (i.e. tumor, metabolic diseases, rheumatoid arthritis, osteoporosis, prolonged history of steroid use, signs and symptoms of vertebrobasilar insufficiency, etc.), use of blood thinners, whiplash injury in the past 6 weeks, evidence of central nervous system involvement (such as hyperreflexia, sensory disturbances in the hands, unsteadiness during walking, etc.), history of spinal surgery, workers compensation or pending legal action regarding their neck pain, insufficient English language skills to complete questionnaires, unable to comply with schedule

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2011-11; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Change in Neck Disability Index (NDI) | baseline; 36-48 hours; 96 hours
  A functional questionnaire completed by the subject

SECONDARY OUTCOMES:
Change in Numeric Pain Rating Scale (NPRS) | baseline; 36-48 hours; 96 hours
Change in Self Reported Activity Scale (SAA) | Baseline; 36-48 hours; 96 hours
Change in Pressure Pain Threshold (PPT) | Baseline; Immediate post intervention; 36-48 hours; 96 hours
Change in Vibratory Measure | Baseline; Immediate post intervention; 36-48 hours; 96 hours
  A specialized tool is used to measure sensory threshold; it is a hand-held sensor with a small vibrating tip held against the skin.
  This device measures how the nerves react to vibration. The procedure is non-invasive. Little or no discomfort should be felt during the test.

OTHER OUTCOMES:
Change in Tampa Scale for Kinesiophobia | Baseline; 36-48 hours; 96 hours
Change in Leeds Assessment of Neuropathic Symptoms and Signs (LANSS) | Baseline; 36-48 hours; 96 hours
Clinical Equipoise | Baseline
  Equipoise occurs when a given treatment has no evidence of being better than another and/or when the individual clinician has no preference of one treatment versus the other.Examiners will complete a form using an 11-point scale to quantify how much they believe the experimental group will have better outcomes or the control group will have better outcomes.
Change in Global Rating of Change (GROC) | Baseline; 36-48 hours; 96 hours
Compliance Measure | 96 hours
  Each patient will complete a daily exercise diary. The examiner will assign a score for compliance based on the patient's knowledge and proficiency of performing their home program and the information in the daily exercise diary.
Change in Range of Motion (ROM) | Baseline; Immediate post intervention; 36-48 hours; 96 hours
Change in Strength | Baseline; immediate post intervention; 36-48 hours; 96 hours

CONTACTS AND LOCATIONS:
Overall Officials: Shannon Petersen, DScPT, Principal Investigator — Des Moines University
Locations (3):
- United States (3):
  - Des Moines University, Des Moines, Iowa
  - Walsh University, North Canton, Ohio
  - Youngstown State University, Youngstown, Ohio